CLINICAL TRIAL: NCT01028326
Title: Immunogenicity and Reactogenicity of 10-valent Pneumococcal Conjugate Vaccine (PCV10) in Children Aged 12-59 Months
Brief Title: PCV10 Reactogenicity and Immunogenicity Study - Malindi
Acronym: PRISM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Collaborators: Kenya Ministry of Health (Other Government); University of Oxford (Other); University of Colorado, Denver (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SSC 1635
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2017-07

CONDITIONS: Pneumococcal Pneumonia
Keywords: Pneumococcal pneumonia vaccine
MeSH Terms: conditions — Pneumonia, Pneumococcal | interventions — 10-valent pneumococcal conjugate vaccine; PHiD-CV vaccine; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Group A of children will receive 2 doses of PCV10 vaccine, one at the time of enrolment and one 2 months later, followed by a dose of DTaP vaccine 4 months later
  Interventions: Biological: PCV10 and DTaP
- Group B (Experimental): Group B of children will receive PCV10 vaccine, followed by a dose of DTaP vaccine after 2 months, and another dose of PCV10 4 months later.
  Interventions: Biological: PCV10 and DTaP
- Group C (Active Comparator): Group C of children will receive a dose of hepatitis A vaccine, followed by a dose of DTaP vaccine after 2 months, and another dose of hepatitis A 4 months later, along with a dose of PCV10.
  Interventions: Biological: hepatitis A vaccine, DTaP, PCV10

INTERVENTIONS:
Biological: PCV10 and DTaP — A nurse will administer a 0.5mL intramuscular dose of PCV10 on day 0 and day 60 and a 0.5 mL intramuscular dose of DTaP on day 180.
  Other Names: Synflorix
  Arms: Group A
Biological: PCV10 and DTaP — A nurse will administer a 0.5mL intramuscular dose of PCV10 on day 0 and day 180 and a 0.5 mL dose of DTaP on day 60.
  Other Names: Synflorix
  Arms: Group B
Biological: hepatitis A vaccine, DTaP, PCV10 — A nurse will administer a 0.5mL intramuscular dose of hepatitis A vaccine on day 0 and day 180; a 0.5 mL intramuscular dose of DTaP on day 60; and a 0.5 mL dose of PCV10 on day 180.
  Other Names: Synflorix
  Arms: Group C

SUMMARY:
The World Health Organization has recommended that developing countries should incorporate pneumococcal conjugate vaccine (PCV) into their routine immunization schedules. The Kenya Ministry of Health anticipates introducing a new formulation of PCV, PCV10, into the routine childhood immunization schedule in 2010. In the areas of Kenya that have been designated to monitor the impact of vaccine, a catch-up campaign will be implemented to vaccinate children aged 12-59 months. PCV10 has been found to be safe and effective in infants. It is licensed for use in children up to 2 years of age, but its use as a primary series in children over age 12 months has not been evaluated. This study will assess the immunogenicity and reactogenicity of PCV10 first administered at an age of 12-59 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-59 months
* Written informed consent

Exclusion Criteria:

* Current febrile illness (temperature >38.5°C)
* Previous receipt of any pneumococcal vaccine
* Previous receipt of a DTP-containing vaccine after the 1st year of life
* Previous receipt of hepatitis A vaccine
* Severe malnutrition (mid upper arm circumference <11.5 cm) or other serious medical condition (e.g., malignancy, AIDS, tuberculosis)
* Seizures within the previous 6 months or progressive neurological illness
* Known allergies to vaccines or vaccine components
* Resident in the Kilifi Demographic Surveillance area
* Intention to leave the study area in the next 6 months

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Serotype-specific anti-pneumococcal antibody responses to vaccination | Day 0, 30, 90, 210

SECONDARY OUTCOMES:
Serotype-specific NP carriage of pneumococci | Day 0, 30, 60, 90, 180
Vaccine reactogenicity | Day 0, 3
Immunological memory responses | Day 0, 30, 90, 210

CONTACTS AND LOCATIONS:
Overall Officials: Laura Hammitt, MD, Principal Investigator — Oxford University, KEMRI-Wellcome Trust
Locations (1):
- Malindi District Hospital, Malindi, Coast, Kenya

REFERENCES:
- [Derived] Feazel LM, Santorico SA, Robertson CE, Bashraheil M, Scott JA, Frank DN, Hammitt LL. Effects of Vaccination with 10-Valent Pneumococcal Non-Typeable Haemophilus influenza Protein D Conjugate Vaccine (PHiD-CV) on the Nasopharyngeal Microbiome of Kenyan Toddlers. PLoS One. 2015 Jun 17;10(6):e0128064. doi: 10.1371/journal.pone.0128064. eCollection 2015. PMID 26083474
- [Derived] Hammitt LL, Ojal J, Bashraheil M, Morpeth SC, Karani A, Habib A, Borys D, Goldblatt D, Scott JA. Immunogenicity, impact on carriage and reactogenicity of 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine in Kenyan children aged 1-4 years: a randomized controlled trial. PLoS One. 2014 Jan 21;9(1):e85459. doi: 10.1371/journal.pone.0085459. eCollection 2014. PMID 24465570